CLINICAL TRIAL: NCT01727414
Title: Medication Response in Children With Predominately Inattentive Type ADHD
Brief Title: Attention Deficit Disorder Medication Response Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADDMedStudy; K23MH083881 (NIH)
Record Dates: First submitted 2012-08-01; First posted 2012-11-16 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: ADHD - Inattentive Type; ADHD - Combined Type
Keywords: ADHD; Inattention; Methylphenidate; Pharmacogenetics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: Every participant receives placebo and three different dose of MPH for one week each in a triple blinded fashion
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OROS-Methylphenidate and placebo for inattentive type pts (Other): Children with ADHD-inattentive type. Every participant receives low dose MPH, medium dose MPH, high dose MPH, and placebo for one week each in a triple-blinded fashion.
  Interventions: Drug: OROS-Methylphenidate and placebo for inattentive type pts
- OROS-Methylphenidate and placebo for combined type pts (Other): Children with ADHD-combined type type. Every participant receives low dose MPH, medium dose MPH, high dose MPH, and placebo for one week each in a triple-blinded fashion.
  Interventions: Drug: OROS-Methylphenidate and placebo for combined type pts

INTERVENTIONS:
Drug: OROS-Methylphenidate and placebo for inattentive type pts — Every participant receives low dose MPH, medium dose MPH, high dose MPH, and placebo for one week each in a triple-blinded fashion.
  Other Names: concerta
  Arms: OROS-Methylphenidate and placebo for inattentive type pts
Drug: OROS-Methylphenidate and placebo for combined type pts — Every participant receives low dose MPH, medium dose MPH, high dose MPH, and placebo for one week each in a triple-blinded fashion.
  Arms: OROS-Methylphenidate and placebo for combined type pts

SUMMARY:
This study evaluates how children with Attention Deficit Disorder without Hyperactivity (ADD) respond to medication, and if their response is different from children who have problems with both hyperactivity and inattention. In order to do this, children ages 7-11 whose primary difficulty is with attention problems and who have never been on behavioral or psychiatric medications are being recruited. Once enrolled, children will try one week each of 3 different doses of methylphenidate, the most commonly prescribed Attention Deficit, Hyperactivity Disorder (ADHD) medication, as well as placebo. Children will be randomly assigned to one of six possible medication dose and placebo titration schedules, but the study doctor, family, and teacher will not know which dose (if any) children are receiving for a given week. Each week, behavioral and side effect ratings will be completed by both the child's parent and teacher, and the family will meet with the study doctor for a physical examination and to discuss how each week went. Some children will also have neuropsychological testing to determine how methylphenidate influences their working memory, sustained attention, and ability to inhibit (stop) inappropriate responses.

All data will be analyzed to decide which medication dose the child responded to best and further recommendations for treatment will be given. Ultimately, this study aims to improve understanding of how children with ADHD-Primarily Inattentive Type respond to stimulant medications by

* determining whether these children experience a diminished response to methylphenidate compared to children with both hyperactivity and inattention
* determining whether certain genetic and environmental factors play a role in this response.

Findings from this study will be used to help streamline the identification of the most effective doses of medication for children with ADHD-Primarily Inattentive Type.

DETAILED DESCRIPTION:
Robust data indicate that stimulant medications reduce ADHD symptoms and impairment, but it is unclear whether their efficacy generalizes across the ADHD subtypes. Although predominately inattentive type (PIT) is the most prevalent ADHD subtype in U.S. population-based studies, few studies have specifically examined response to stimulants in this subtype. Instead, medication guidelines for PIT have largely been extrapolated from studies enrolling all or mostly ADHD-combined type (CT). Thus, this application seeks to improve understanding of stimulant medication response and its predictors in children with PIT. We will evaluate participants' response to methylphenidate (MPH), the most widely prescribed stimulant, via a prospective, double-blind, placebo-controlled crossover trial with 3 dose conditions. Our first specific aim is to examine MPH medication and dose response in children with PIT (n=120) and CT (n=45) to test the hypotheses that participants with PIT have a diminished MPH response and derive less benefit from higher doses compared to those with CT. Since only one prior study has examined genetic predictors of MPH response variability within PIT-only samples, our second specific aim (exploratory) is to determine the potential role of genetic polymorphisms (e.g., those in DAT1, DRD4, NET, ADRA2A, COMT, SNAP25, CES1, GRM7, LPHN3) on MPH response in children with PIT (n=120), examining both symptom change with MPH and MPH dose response curves. If we identify significant differences in MPH response between the subtypes, our findings may guide clinical practice by suggesting more effective medication strategies (such as different dosing schedules) for children with PIT. In addition, this study may yield pharmacogenetic findings that, in the future, could enable physicians to tailor individual treatment plans for children with PIT, ameliorating the current prolonged and expensive practice of prescribing by trial and error.

ELIGIBILITY:
Inclusion Criteria:

* Consent: The family must provide signature of informed consent by a parent or legal guardian. Children must also assent to study participation.
* Age at Screening:7.0 years to 11.9 years, inclusive.
* Sex: Includes male and female children.
* ADHD Diagnostic Status: Meets DSM-IV criteria for ADHD, Predominantly Inattentive or Combined subtype with Clinical Global Impression-Severity rating corresponding to at least "moderately ill."
* Cognitive Functioning-Intelligence Quotient (IQ) of greater than 80 as estimated by Vocabulary and Block Design subtests of the Wechsler Intelligence Scale for Children--4th Edition, or an Intelligence Quotient (IQ) of 80 or greater when administered the Full Scale Version of the Wechsler Intelligence Scale for Children-4th Edition.
* Absence of Learning Disability:On the abbreviated Wechsler Individual Achievement Test-2nd edition Reading and Math subtests, participants must score above 80. However, children may also be included if they receive a score of 75 or greater on the Word Reading and/or Math subtests, as long as this score is not a significant discrepancy from their full-scale IQ score (e.g., a difference of greater than one standard deviation or 15 points).
* School: Enrolled in a school setting rather than a home-school program.

Exclusion Criteria:

* Understanding Level: Participant and/or parent cannot understand or follow study instructions.
* Psychiatric Medications: Current or prior history of taking any medication for psychological or psychiatric problems.
* Behavioral Interventions: Current active participation in ADHD-related behavioral interventions or counseling.
* Exclusionary Psychiatric Conditions: Children with mania/hypomania and/or schizophrenia will be excluded. The following comorbid diagnoses will not be excluded unless they are determined to be the primary cause of ADHD symptomatology (see below for description of this decision process): Post Traumatic Stress Disorder, Phobias and Anxiety Disorders, Obsessive Compulsive Disorder, Major Depression / Dysthymia, Eating Disorders, Elimination Disorders, Trichotillomania, Tic Disorder, Oppositional Defiant Disorder, Conduct Disorder.
* Organic Brain Injury: History of head trauma, neurological disorder, or other organic disorder affecting brain function.
* Cardiovascular Risk Factors: Children with a personal history or family history of cardiovascular risk factors will be excluded, or given the option of participating in the study after obtaining an EKG and a signed letter from a pediatric cardiologist verifying the safety of their participation in a trial of methylphenidate. In this case, families will be responsible for the costs of EKG and cardiologist evaluation. If for any reason a family is unable to assume the cost of the EKG and cardiologist evaluations but still wishes for their child to participate, study staff will determine on a case-by-case basis whether the study budget allows the study to offer financial assistance to the families for these evaluations.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2006-06; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya E. Froehlich, MS, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Froehlich TE, Becker SP, Nick TG, Brinkman WB, Stein MA, Peugh J, Epstein JN. Sluggish Cognitive Tempo as a Possible Predictor of Methylphenidate Response in Children With ADHD: A Randomized Controlled Trial. J Clin Psychiatry. 2018 Mar/Apr;79(2):17m11553. doi: 10.4088/JCP.17m11553. PMID 29489078

RESULTS

PARTICIPANT FLOW:
Groups:
- Inattentive Type: Every participant receives low dose MPH, medium dose MPH, high dose MPH, and placebo for one week each in a triple-blinded fashion.
  Placebo: capsule, frequency - each AM, duration - 1 week
- Combined Type: Every participant receives low dose MPH, medium dose MPH, high dose MPH, and placebo for one week each in a triple-blinded fashion.
  OROS-Methylphenidate: capsule; dosages - 18mg, 27mg, 36mg, 54 mg; frequency - each AM; duration - one week for each dose, with each child receiving 3 doses [children < 25 kg receive 18mg, 27mg, 36mg; children > or = to 25kg get 18mg, 36mg, 54mg]
Period: Overall Study
Arm/Group | Inattentive Type | Combined Type
Started | 126 | 45
Completed | 123 | 45
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Children meeting DSM-IV criteria for ADHD-inattentive type are in the Inattentive Type Arm, while children meeting DSM-IV criteria for ADHD-combined type are in the Combined Type Arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Inattentive Type | Combined Type | Total
Number analyzed (Participants) | 126 | 45 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (1.3) | 7.9 (1.0) | 8.4 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 9 | 49
  Male | 86 | 36 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 15 | 21
  White | 109 | 30 | 139
  More than one race | 8 | 0 | 8
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Attention Deficit Hyperactivity Disorder Total Symptom Score
Description: Assessed via parent and teacher Vanderbilt Attention Deficit Hyperactivity Disorder Rating Scales which were completed each the 4 weeks of the titration trial.
  Range: min=0, max=54 [sum of 18 symptom items, rated from 0 (none), 1 (occasionally), 2 (often), 3 (very often)], higher scores indicate worse outcomes.
  Note to address Review Comment: During the 4 week titration trial, the placebo condition and each of the three active dosages (low, medium, and high) were given for one week each. Because the placebo and active dosages were given in random order to preserve the triple blind, all participants did not receive the same order of dosages and it is not possible to connect the dosages (placebo, low dose MPH, medium dose MPH, high dose MPH) to a specific week number (week 1, week 2, week 3, week 4) which would hold for ALL participants. That is why Timeframe was revised from "week 1, week 2, week 3, week 4" to placebo, low dose, medium dose, and high dose week.
Time Frame: End of placebo dose week, End of low dose week, End of medium dose week , End of high dose week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Inattentive Type; Combined Type: Every participant receives low dose MPH, medium dose MPH, high dose MPH, and placebo for one week each in a triple-blinded fashion.
  OROS-Methylphenidate: capsule; dosages - 18mg, 27mg, 36mg, 54 mg; frequency - each AM; duration - one week for each dose, with each child receiving 3 doses [children < 25 kg receive 18mg, 27mg, 36mg; children > or = to 25kg get 18mg, 36mg, 54mg]
Arm/Group | Inattentive Type | Combined Type
Number analyzed (Participants) | 123 | 45
units on a scale
  ADHD Total Symptom Score on Placebo | 21.4 (8.9) | 30.0 (9.2)
  ADHD Total Symptom Score on Low Dose MPH | 20.2 (8.1) | 29.7 (10.6)
  ADHD Total Symptom Score on Medium Dose MPH | 17.0 (7.9) | 23.9 (10.7)
  ADHD Total Symptom Score on High Dose MPH | 15.5 (6.9) | 22.8 (10.8)
Statistical Analysis 1: Comparison: Inattentive Type vs Combined Type; Test type: Superiority — General linear mixed models were used to evaluate the subtype*dose interaction to determine if the subtypes have unique MPH dose-response curves, with the outcome being Attention Deficit Hyperactivity Disorder total symptom scores (minimum=0, maximum=54, higher=worse); p < 0.05, Mixed Models Analysis; Slope = 0.29

ADVERSE EVENTS:
Time Frame: 4 week medication titration trial
Groups:
- Inattentive Type: Children meeting DSM-IV criteria for ADHD-inattentive type.
- Combined Type: Children meeting DSM-IV criteria for ADHD-combined type.
Arm/Group | Inattentive Type | Combined Type
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/45
Other Adverse Events (participants affected / at risk) | 17/123 | 8/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inattentive Type (N=123) | Combined Type (N=45)
Irritability (Nervous system disorders) | 17 (17) | 8 (8) — Parent rating of having moderate or severe irritability on the Pittsburgh side effect rating scale while taking the highest methylphenidate dose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No